CLINICAL TRIAL: NCT06829472
Title: Conditioning Regimen of Melphalan-busulfan and Fludarabine: a Randomize Study Comparing 100mg/m2 to 140mg/m2 Melphalan for Adult Patients With Acute Myeloid Leukemia or Myelodysplasia Syndrome.
Brief Title: Conditioning Regimen of Melphalan-busulfan and Fludarabine: a Randomized Study of Different Dose of Melphalan
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Clinical Research Center (Unknown)
Responsible Party: Principal Investigator, Jiong HU, Deputy director, Department of Hematology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBF-RJH-2023
Record Dates: First submitted 2023-08-12; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Toxicities; Survivorship
Keywords: melphalan, AML, MDS, allogeneic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Melphalan

STUDY DESIGN:
Intervention Model Description: Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBF100 (Experimental): Patients receive condoning regimen with melphalan (100mg/m2) with busulfan and fludarabine.
  Interventions: Drug: melphalan
- MBF140 (Active Comparator): Patients receive condoning regimen with melphalan (140mg/m2) with busulfan and fludarabine.
  Interventions: Drug: melphalan

INTERVENTIONS:
Drug: melphalan — conditioning regimen with melphalan, busulfan and fludarabine
  Other Names: MBF

SUMMARY:
Conditioning regimen with melphalan-busulfan and fludarabine (MBF) achieved low relapse rate in patients with acute myeloid leukemia (AML) and myelodysplasia syndrome (MDS). In our previous retrospective study, we demonstrated that melphalan dose at 100 or 140mg/m2 had similar incidence of relapse but it might had lower toxicities. In this prospective randomize study, we aim to compare the transplantation outcome in adult patients with AML/MDS receiving either MBF with 100 or 140 mg/m2 melphalan.

DETAILED DESCRIPTION:
Intensity of conditioning regimen plays a important role in allogeneic stem cell transplantation (allo-HSCT) for patents with AML and MDS. IN our previous prospective study, we demonstrated that condoning regimen of dual alkylating agents with melphalan-busulfan and fludarabine (MBF) achieved a very low relapse rate (~6%) in patients with acute myeloid leukemia (AML) and myelodysplasia syndrome (MDS). In that study, adult patients received melphalan 140mg/m2 while patients >=60 or with high transplantation risk in terms of HCT-CI received reduced dose of melphalan (100mg/m2). Overall, it was shown that 100 or 140mg/m2 melphalan had similar incidence of relapse while the 100mg/m2 melphalan presented lower incidence of toxicities.In this prospective randomize study, we aim to compare the transplantation toxicities and outcomes in young adults (18~55) with AML/MDS receiving either 100 or 140 mg/m2 melphalan as conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML in first remission
* Patients with MDS with bone marrow blast >5% but remain less than 20% before transplantation
* Donor available: HLA matched sibling donor, 9~10/10 matched unrelated donor or haplo-identical donor
* Inform consent provided

Exclusion Criteria:

* Patients with active infection (bacteria, fungal or viral)
* Patients with abnormal liver, renal and cardiac function

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Toxicities | up to 100 days
  Toxicities with grade III or over

SECONDARY OUTCOMES:
Relapse | 2 years
  Documentation of bone marrow blasts >5% or extra medullary disease
Non-relapse mortality | 100 days
  Death without documentation of AML and MDS disease
Non-relapse mortality | 2 years
  Death without documentation of AML and MDS disease
disease-free survival | 2 years
  event defined as documentation of AML and MDS relapse or death of any causes
overall survival | 2 years
  event defined as death of any causes

CONTACTS AND LOCATIONS:
Overall Officials: chun Wang, Study Director — Go Broad Health Care
Locations (2):
- China (2):
  - Rui Jin Hospital, Shanghai, Shanghai Municipality
  - Zhaxin Hospital, Go Broad Health Care, Shanghai, Shanghai Municipality